CLINICAL TRIAL: NCT05546333
Title: Assessing the Effectiveness of Electrical Impedance Tomography Images to Detect Pulmonary Emboli Compared to Computed Tomographic Angiography
Brief Title: Comparing Electrical Impedance Tomography to Computed Tomographic Angiography
Status: Active, not recruiting | Type: Observational
Sponsor: Colorado State University (Other)
Collaborators: UC Health Medical Center of the Rockies (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21-4600
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving CTA: Patients who will receive a CTA due to clinical need will be imaged with electrical impedance tomography in addition to the CTA.
  Interventions: Device: Electrical impedance tomography

INTERVENTIONS:
Device: Electrical impedance tomography — Non-invasive measure of electrical impedance in the body, with data collected on electrodes on the surface of the body
  Other Names: EIT

SUMMARY:
The study aim is to determine whether electrical impedance tomography (EIT) is equivalent in the detection of pulmomary emboli compared to Computed Tomographic Angiography (CTA). EIT is a non-invasive, non-ionizing functional imaging technique that can be performed at bedside. Electrical impedance tomography data will be collected on individuals undergoing a CTA scan of the chest at Medical Center of the Rockies (MCR). The primary outcome measure is to assess whether assessment by CTA corresponds with EIT in detection of pulmonary emboli. The study will include up to 63 participants. EIT data will be collected for up to 20 minutes during tidal breathing and for approximately five to ten seconds during breath-holding.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing a CTA of the chest at MCR

Exclusion Criteria:

* Under 18 years of age
* Body mass index (BMI) > 30
* Individuals with known thoracic metal implants or devices, such as pacemakers (internal and external), staples, or spinal and rib hardware
* Individuals deemed by the research team as too unstable to safely apply the EIT belt, such as hemodynamic or respiratory instability (e.g., intubated patients), and individuals with unstable spinal injuries
* Open wounds at the site of electrode belt application

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals undergoing a CTA scan of the chest at Medical Center of the Rockies (MCR) for a suspected pulmonary embolism
Sampling Method: Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
Correspondence to CTA | One year
  To assess whether assessment by CTA corresponds with EIT in detection of pulmonary emboli (PE).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Mueller, PhD, Principal Investigator — Colorado State University
Locations (1):
- UCHealth Medical Center of the Rockies, Loveland, Colorado, United States

IPD SHARING:
Plan to Share IPD: No